CLINICAL TRIAL: NCT03965494
Title: Pilot Surgical PK Study of BGB324 in Recurrent Glioblastoma Patients
Brief Title: AXL Inhibitor BGB324 in Treating Participants With Recurrent Glioblastoma Undergoing Surgery
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: NCI decided to terminate ABTC Consortium due to NCI moving in different direction for Brain Cancer - official close date is 10/31/23
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH); BerGenBio ASA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABTC-1701; IRB00184546 (Other: JHM IRB); UM1CA137443 (NIH)
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma | interventions — bemcentinib; Postoperative Period

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AXL inhibitor BGB324 then surgery (Experimental): Participants receive AXL inhibitor BGB324 PO QD on days 1-5, then undergo surgery 3-6 hours after last dose. Within 45 days, participants receive AXL inhibitor BGB324 PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: BGB 324 (before surgery)
- Surgery then AXL inhibitor BGB324 (Experimental): Participants undergo surgery, then within 45 days receive AXL inhibitor BGB324 PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: BGB 324 (after surgery)

INTERVENTIONS:
Drug: BGB 324 (before surgery) — Given by mouth either BEFORE therapeutic conventional surgery
  Other Names: AXL Inhibitor BGB324; Bemcentinib
  Arms: AXL inhibitor BGB324 then surgery
Drug: BGB 324 (after surgery) — Given by mouth either AFTER therapeutic conventional surgery
  Other Names: AXL Inhibitor BGB324; Bemcentinib
  Arms: Surgery then AXL inhibitor BGB324

SUMMARY:
This phase I trial studies how well AXL inhibitor BGB324 works in treating participants with glioblastoma that has come back who are undergoing surgery. AXL inhibitor BGB324 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the penetration of AXL inhibitor BGB324 (BGB324) across the blood brain barrier measured by pharmacokinetics/drug concentration of 1.0 uM in tissue resected from a contrast enhancing region of the tumor in 60% of recurrent glioblastoma patients.

SECONDARY OBJECTIVES:

I. Determine AXL expression, phosphorylation state (AXL phosphospecific antibody if AXL is inhibited), and circulating soluble AXL levels.

II. Determine the BGB324 concentration in tissue resected from a contrast non-enhancing region of the tumor.

III. Characterize the steady state pharmacokinetics of BGB324 in patients with recurrent glioblastoma.

IV. Estimate safety and tolerability of BGB324 for recurrent glioblastoma. V. Assess the progression-free and overall survival of patients with recurrent glioblastoma.

OUTLINE: Participants are assigned to 1 of 2 groups.

GROUP A: Participants receive AXL inhibitor BGB324 orally (PO) once daily (QD) on days 1-5, then undergo surgery 3-6 hours after last dose. Within 45 days, participants receive AXL inhibitor BGB324 PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

GROUP B: Participants undergo surgery, then within 45 days receive AXL inhibitor BGB324 PO QD on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically confirmed glioblastoma (GBM) that is progressive or recurrent following radiation therapy +/- chemotherapy. Patients with previous low-grade glioma who progressed after radiation therapy (RT)/chemotherapy and are biopsied and found to have GBM/gliosarcoma (GS) are eligible
* Patients must have measurable, supratentorial contrast-enhancing progressive or recurrent glioblastoma or gliosarcoma by magnetic resonance imaging (MRI) within 21 days of starting treatment. Patient must be able to tolerate MRIs
* May have had treatment for no more than 2 prior relapses
* Must have a tumor tissue form indicating availability of archived tissue from initial resection at diagnosis of GBM or GS, completed and signed by a pathologist. Sites must agree to provide this form within 14 days after treatment start. Availability of tissue is not a requirement for study participation
* The following intervals from previous treatments are required to be eligible:

  * 12 weeks from the completion of radiation
  * 6 weeks from a nitrosourea chemotherapy or mitomycin C
  * 3 weeks from a non-nitrosourea chemotherapy
  * 4 weeks from any investigational (not Food and Drug Administration [FDA]-approved) agents
  * 2 weeks from administration of a non-cytotoxic, FDA-approved agent, e.g., erlotinib, hydroxychloroquine, etc.)
  * 4 weeks from prior antiangiogenesis therapy (approved or investigational) (e.g., bevacizumab, aflibercept, ramucirumab, cediranib, cabozantinib, etc.)
  * 4 weeks from any immunotherapy intervention
* Patients must be undergoing surgery that is clinically indicated as determined by their care providers. Patients must be eligible for surgical resection according to the following criteria:

  * Expectation that the surgeon is able to resect 0.05-0.10 cm^3 (50-100 mg) of tumor from enhancing tumor and at least 0.05-0.10 cm^3 (50-100 mg) from non-enhancing tumor with low risk of inducing neurological injury
* Must have a Karnofsky performance status >= 60% (i.e. the patient must be able to care for himself/herself with occasional help from others)
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Hemoglobin >= 9 g/dL
* Total bilirubin < 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 x institutional upper limit of normal
* Creatinine =< institutional upper limit of normal OR creatinine clearance >= 60 ml/min/1.73m^2 for patients with creatinine levels above institutional normal
* Activated partial thromboplastin time (APTT)/partial thromboplastin time (PTT) =< 1.5 x institutional upper limit of normal
* Must have a 12-lead electrocardiogram with a measurable corrected QT using Fridericia's correction formula (QTcF) =< 450 msec
* Must be able to provide written informed consent
* Women of childbearing potential must have a negative serum pregnancy test prior to study entry. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, and through 4 months after the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of BGB324 administration
* Must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder. Patients with prior malignancies must be disease-free for >= five years
* Must be able to swallow whole capsules

Exclusion Criteria:

* Patients receiving any other investigational agents are ineligible
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to BGB324 are ineligible. The investigator brochure can be referenced for more information
* Patients on enzyme-inducing anti-epileptic drugs (EIAED) are not eligible for treatment on this protocol. Patients may be on non-enzyme inducing anti-epileptic drugs or not be taking any anti-epileptic drugs. Patients previously treated with an EIAED may be enrolled if they have been off the EIAED for 10 days or more prior to treatment start
* Patients with a history of bleeding diathesis are ineligible
* Patients who have not recovered to < Common Terminology Criteria for Adverse Events (CTCAE) grade 2 toxicities related to prior therapy are ineligible
* Patients considered at risk of QTc induced arrhythmias or uncontrolled or significant cardiovascular disease, including, but not limited to, any of the following are ineligible:

  * Abnormal left ventricular ejection fraction on echocardiography (less than the lower limit of normal for a subject of that age at the treating institution or < 45%)
  * History of an ischemic cardiac event including myocardial infarction within 3 months of study entry
  * Congestive cardiac failure of > grade 2 severity according to the New York Heart Association as defined by symptomatic at less than ordinary levels of activity
  * Unstable cardiac disease including unstable angina or hypertension as defined by the need for change in medication within the last 3 months
  * History or presence of bradycardia (=< 60 beats per minute [bpm]) or history of symptomatic bradycardia, left bundle branch block, cardiac pacemaker or significant atrial tachyarrhythmias as defined by the need for treatment
  * Current treatment with any agent known to cause torsade de points which cannot be discontinued at least two weeks prior to treatment
  * Known family or personal history of long QTc syndrome or ventricular arrhythmias including ventricular bigeminy
  * Previous history of drug-induced QTc prolongation
  * Screening 12-lead electrocardiogram (ECG) with a measurable QTcF > 450 ms
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, clinically significant cardiac disease, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, are ineligible
* Pregnant women are excluded from this study because the effects of BGB324 on a fetus are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with BGB324, breastfeeding should be discontinued if the mother is treated with BGB324
* Patients positive for human immunodeficiency virus (HIV) are NOT excluded from this study, but HIV-positive patients must have:

  * A stable regimen of highly active anti-retroviral therapy (HAART) not containing a strong inducer or inhibitor of CYP2C9
  * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
  * A CD4 count above 250 cells/uL and an undetectable HIV viral load on standard polymerase chain reaction (PCR)-based test

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who achieve a drug concentration at >= 1.0 uM level in contrast enhancing tumor tissue | Up to 1 year
  Will be estimated using binomial distribution along with 90% confidence interval.

SECONDARY OUTCOMES:
Change in AXL expression level | Up to 1 year
  Change in AXL expression level (ng/mL) from baseline (before intervention) to post-intervention.
Pharmacokinetics as measured by plasma maximum concentration (Cmax) (ug/mL) | up to 30 days post-treatment
  Samples for pharmacokinetic analysis will be collected at baseline, prior to dose on day of surgery, at 2, 4, 8, 12, 16, 20, and 24 hours after dosing; on course (C)1 day (D)1, at 2, 4, 6 and 24 hours on C1D15, C2D8, C2D15, prior to starting each course and 30 days post-treatment
Pharmacokinetics as measured by plasma minimum concentration (Cmin) (ug/mL) | up to 30 days post-treatment
  Samples for pharmacokinetic analysis will be collected at baseline, prior to dose on day of surgery, at 2, 4, 8, 12, 16, 20, and 24 hours after dosing; on course (C)1 day (D)1, at 2, 4, 6 and 24 hours on C1D15, C2D8, C2D15, prior to starting each course and 30 days post-treatment
Pharmacokinetics as measured by area under the curve (AUC) (ug/mL*hr) | up to 30 days post-treatment
  Samples for pharmacokinetic analysis will be collected at baseline, prior to dose on day of surgery, at 2, 4, 8, 12, 16, 20, and 24 hours after dosing; on course (C)1 day (D)1, at 2, 4, 6 and 24 hours on C1D15, C2D8, C2D15, prior to starting each course and 30 days post-treatment
Toxicity as assessed by number of participants experiencing of adverse events | Up to 1 year
  Number of participants experiencing of adverse events grade 3 or higher as defined by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v5.0)
Overall survival | up to 1 year
  Time until death or the time of last known alive if lost to follow-up. Survival probability and a median time of survival will be estimated using Kaplan-Meier method along with 95% confidence interval.
Progression-free survival | up to 1 year
  Median time of progression-free survival will be estimated using Kaplan-Meier method along with 95% confidence interval. Tumor assessment will be conducted per Response Assessment in Neuro-Oncology (RANO): Complete Response (CR)= no change in size of T1-gadolinium-enhancing (T1-Gd+) disease, stable or reduced T2/FLAIR signal, no new lesion, no corticosteroid use, and stable or improved clinical status; Partial Response (PR)= ≥50% change in size of T1-Gd+ disease, stable or reduced T2/FLAIR signal, no new lesion, stable or reduced corticosteroid use, and stable or improved clinical status; Stable Disease (SD)= <50% reduction to <25% increase size of T1-Gd+ disease, stable or reduced T2/FLAIR signal, no new lesion, stable or reduced corticosteroid use, and stable or improved clinical status; Progressive Disease (PD)= ≥25% increase size of T1-Gd+ disease, or increased T2/FLAIR signal, or presence of new lesion, or worsening clinical status

CONTACTS AND LOCATIONS:
Overall Officials: Burt Nabors, MD, Study Chair — University of Alabama and Birmingham
Locations (6):
- United States (6):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Memorial Sloan Kettering, New York, New York
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No